CLINICAL TRIAL: NCT06452225
Title: Ultrasound Guided Transversus Abdominis Plane Block Versus External Oblique Intercostal Plane Block for Postoperative Analgesia in Pediatrics Undergoing Open Nephrectomy
Brief Title: Transversus Abdominis Plane Block Versus External Oblique Intercostal Plane Block for Postoperative Analgesia in Pediatrics Undergoing Open Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR641/4/24
Record Dates: First submitted 2024-05-30; First posted 2024-06-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Transversus Abdominis Plane Block; External Oblique Intercostal Plane Block; Postoperative Analgesia; Pediatrics; Open Nephrectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External Oblique Intercostal Plane Block (Experimental): Patients will receive external oblique intercostal plane block.
  Interventions: Other: External Oblique Intercostal Plane Block
- Transversus Abdominis Plane Block (Experimental): Patients will receive ultrasound guided transversus abdominis plane block.
  Interventions: Other: Transversus Abdominis Plane Block

INTERVENTIONS:
Other: External Oblique Intercostal Plane Block — Patients will receive external oblique intercostal plane block.
  Arms: External Oblique Intercostal Plane Block
Other: Transversus Abdominis Plane Block — Patients will receive ultrasound guided transversus abdominis plane block.
  Arms: Transversus Abdominis Plane Block

SUMMARY:
The aim of this study is to compare the ultrasound guided TAP Block and EOIP block for postoperative analgesia in pediatrics undergoing open nephrectomy.

DETAILED DESCRIPTION:
Nephrectomy in children may also be for malignant conditions of the kidney and adrenal glands. The major indications for nephrectomy vary in different parts of the world and in different age groups and sexes with some recording more benign conditions and others more of malignancies Ultrasound-guided transversus abdominis plane (TAP) block is a relatively new technique to infiltrate regional anesthesia in which local routine anesthetics are injected between the internal oblique and transverse abdominal muscles. The purpose is to provide analgesia to the parietal peritoneum as well as the skin and muscles of the anterior abdominal wall.

External oblique intercostal plane block (EOIPB) has been reported by Elsharkawy et al. in 2021 as a significant modification of fascial plane blocks in that it may engage the upper lateral abdominal walls consistently. In comparison to quadratus lumborum block (QLB) and erector spinae plane block (ESPB) , The advantage of EOIPB is that it may be performed with the patient supine. Furthermore, in comparison to serratus intercostal plane block (SIPB), it generates more extensive analgesic effects throughout the whole midline of the abdomen .

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 18 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-III.
* Scheduled for open nephrectomy.

Exclusion Criteria:

* Abnormal blood coagulation.
* Scar, infection, and tumor of puncture site.
* History or family history of high malignant fever.
* Severe cardiovascular problems.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  A standardized analgesic regimen will be prescribed in the post-operative period. All patients will receive paracetamol 15 mg /kg/8 hrs as routine analgesia. Rescue analgesia of morphine will be given as 0.05 mg/kg if face, legs, activity, and cry consolability scale (FLACC) ≥ 4 and the maximum allowed dose is 0.1mg/kg every 4 hours. FLACC will be assessed at 0, 2, 4, 8, 12 and 24h postoperatively.
  it will be measured from the end of surgery to first dose of morphine administrated.

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | Intraoperatively
  Additional fentanyl bolus dosages of 1 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 0.05 mg/kg if the face, legs, activity, and cry consolability scale (FLACC) ≥ 4 and the maximum allowed dose is 0.1mg/kg every 4 hours.
Degree of pain | 24 hours postoperatively
  The pain will be assessed by using the face, legs, activity, and cry consolability scale (FLACC). The level of response for each observation is given a numerical value rating from "0" to "2," with "0" being the most comfortable with no pain and "2" being the most painful , which results in a total score between "0" and "10".
  It will be assessed at 0, 2, 4, 8, 12 and 24h postoperatively.
Mean arterial pressure | Every 15 minutes till the end of surgery
  Mean arterial pressure will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.

OTHER OUTCOMES:
Heart rate | Every 15 minutes till the end of surgery
  Heart rate will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year
Supporting Information: Study Protocol
Time Frame: After the end of study for one year
Access Criteria: The data will be available upon a reasonable request from the corresponding author